CLINICAL TRIAL: NCT04238962
Title: A Trial to Demonstrate Bioequivalence Between the Semaglutide D Formulation for the DV3396 Pen-Injector and the Formulation for the PDS290 Pen-Injector Following Subcutaneous Administration of 2 mg Semaglutide
Brief Title: A Research Study to Compare Two Different Forms of Once-weekly Semaglutide in Two Different Injection Pens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4601; U1111-1239-1473 (Other: World Health Organization (WHO)); 2019-003477-25 (Registry Identifier: European Medicines Agency (EMA))
Record Dates: First submitted 2020-01-22; First posted 2020-01-23 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DV3396 (Experimental): Participants will receive once-weekly doses of semaglutide administered with the DV3396 pen-injector (test drug product)
  Interventions: Drug: Semaglutide (administered by DV3396 pen-injector)
- PDS290 (Active Comparator): Participants will receive once-weekly doses of semaglutide administered with the PDS290 pen-injector (comparator drug product)
  Interventions: Drug: Semaglutide (administered by PDS290 pen-injector)

INTERVENTIONS:
Drug: Semaglutide (administered by DV3396 pen-injector) — Increasing doses of semaglutide given subcutaneously (sc, under the skin) in the stomach for 7 weeks
  Arms: DV3396
Drug: Semaglutide (administered by PDS290 pen-injector) — Increasing doses of semaglutide given sc in the stomach for 7 weeks
  Arms: PDS290

SUMMARY:
The study will look at how 2 different semaglutide versions reach and stay in the blood after injection. The study aims to show similar levels of semaglutide in the blood when using the different semaglutide versions. Participants will get 1 of the 2 versions of semaglutide - which version is decided by chance. One version is the one that doctors already can prescribe and the other is the new version. Participants will get the medicine as an injection under the skin of the belly with a pen-injector. The type of pen-injector is different for the 2 versions of semaglutide. Participants will receive 7 once-weekly injections in total. The study will last for about 80-106 days. Participants will have 19 study visits with the study doctor. For 2 of the visits, participants will stay in the clinic, 1 visit for 2 days and 1 night and the other visit for 4 days and 3 nights. Participants may have to stop the study if the study doctor thinks that there are risks for their health. Participants cannot take part in this study if they have any disease or disorder that the study doctor thinks is a health problem. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-65 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 25.0 and 34.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Body weight between 65.0 and 130.0 kg (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive methods.
* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.
* Use of prescription medicinal products or non-prescription drugs or herbal products, except routine vitamins, topical medication, highly effective contraceptives and occasional use of paracetamol and acetylsalicylic acid (the two latter are not allowed within 24 hours before screening), within 14 days prior to the day of screening.
* Abuse or intake of alcohol, defined as any of the below:
* Known or suspected alcohol abuse within 1 year prior to the day of screening (defined as regular intake of more than an average intake of 24 g alcohol daily for men and 12 g alcohol daily for women -12 g of alcohol equals about 300 mL of beer or lager, 100 mL of wine, or 25 mL spirits)
* Positive alcohol test at screening
* Abuse or intake of drugs, defined as any of the below:
* Known or suspected drug/chemical substance abuse within 1 year prior to the day of screening
* Positive drug of abuse test at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
AUC0-last,sema,2mg: Area under the semaglutide concentration time curve from time 0 until last quantifiable measurement after one dose of s.c. semaglutide 2 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 2 mg
  h*nmol/L
Cmax,sema,2mg: Maximum observed semaglutide concentration after one dose of s.c. semaglutide 2 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 2 mg
  nmol/L

SECONDARY OUTCOMES:
AUC0-∞,sema,2mg: Area under the semaglutide concentration time curve from time 0 until infinity after one dose of s.c. semaglutide 2 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 2 mg
  h*nmol/L
tmax,sema,2mg: Time of maximum observed semaglutide concentration after one dose of s.c. semaglutide 2 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 2 mg
  h
t½,sema,2mg: terminal elimination half-life of semaglutide after one dose of s.c. semaglutide 2 mg administration following a 6-week dose escalation period | 0-840 hours after one dose of s.c. semaglutide 2 mg
  h

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com